CLINICAL TRIAL: NCT01854606
Title: An Open-Label, Single-arm, Phase Ib/II Study of AEB071 (a Protein Kinase C Inhibitor) and Everolimus (mTOR Inhibitor) in Patients With CD79-mutant or ABC Subtype Diffuse Large B-Cell Lymphoma
Brief Title: Safety and Efficacy of AEB071 and EVEROLIMUS in Patients With CD79-mutant or ABC Subtype Diffuse Large B-Cell Lymphoma
Acronym: COEB071X2103
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COEB071X2103
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-05

CONDITIONS: CD79 Mutant or ABC-subtype Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma, DBCL, AEB071, Everolimus
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — sotrastaurin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AEB071 and EVEROLIMUS (Experimental): AEB071 and EVEROLIMUS will be taken together in this open-label non-randomized study
  Interventions: Drug: AEB071; Drug: Everolimus

INTERVENTIONS:
Drug: AEB071 — a Protein Kinase C Inhibitor
  Other Names: sotrastuarin
Drug: Everolimus — mTOR inhibitor
  Other Names: RAD001

SUMMARY:
Study of the safety and efficacy of AEB071 and EVEROLIMUS in patients with CD79-mutant or ABC subtype Diffuse Large B-Cell Lymphoma.

The trial did not progress into Phase II due to the suboptimal tolerability of the combination treatment of sotrastaurin and everolimus in the Phase Ib part of the study. There were no serious safety concerns associated with this combination.

DETAILED DESCRIPTION:
This is a Phase Ib dose escalation and Phase II study in patients with DLBCL harboring mutations in CD79A/B or of the ABC subtype. Pre-screening for mutations in CD79A/B or the ABC subtype will be required, as it is anticipated that both patient groups may receive clinical benefit from the combination of AEB071 and EVEROLIMUS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Diffuse DLBCL with activating mutations in CD79 (A or B subunits) or ABC-subtype DLBCL (CD79 wildtype or CD79 mutant). DLBCL that arose from transformed indolent lymphoma is allowed.
* Prior treatment and relapse following chemotherapy and autologous bone marrow or stem cell transplant. Patients who are not transplant eligible or who did not respond to chemotherapy may be considered for the study following a single regimen of chemotherapy such as R-CHOP or R-EPOCH. There is no limit to number of prior therapies allowed.
* May be treated with localized radiation as long as measurable or evaluable disease remains at untreated sites.
* WHO performance status of ≤ 2.
* A representative FFPE tumor sample must be available for molecular testing along with a corresponding pathology report. An archival tumor sample may be submitted. However, if not available, a new tumor biopsy obtained for the purpose of this study must be submitted instead.

Exclusion Criteria:

* Treatment with strong inducers or inhibitors (medications and herbal supplements) of cytochrome P450 3A4/5 (CYP3A4/5), or CYP3A4/5 substrates with a QT prolongation risk that cannot be discontinued at least 7 half-lives (or if the half-life is unknown,14 days) prior to study drug treatment.
* Impaired cardiac function or clinically significant cardiac diseases.
* Impairment of GI function or GI disease that could interfere with the absorption of AEB071 or everolimus.
* Severe systemic infections, current or within the two weeks prior to initiation of AEB071.
* Kown history of HIV.
* Poorly controlled diabetes as defined by a fasting serum glucose > 2.0 x ULN.
* Evidence of current CNS involvement.
* Significant symptomatic deterioration of lung function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Phase Ib- Incidence of dose limiting toxicities (DLT) during the first cycle | 12 months
  Estimate the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of the AEB071and EVEROLIMUS combination therapy in patients with DLBCL.
Phase II- Overall response rate (ORR) = complete response (CR) + partial response (PR) according to the non-Hodgkin's Lymphoma International Working Group criteria | 12 months
  Assess the preliminary evidence for anti-tumor activity at RP2D for AEB071 and EVEROLIMUS in patients with a CD79 mutation and those wild-type for the mutation but of the ABC subtype

SECONDARY OUTCOMES:
Occurrence of Adverse Events (AEs), Serious Adverse Events (SAEs) assessments of clinical laboratory values and vital sign measurements. | 24 months
  Safety and tolerability of AEB071 and EVEROLIMUS, including acute and chronic toxicities
Best Overall Response (BOR) | 24 months
  Evaluate preliminary anti-tumor activity for AE071 and EVEROLIMUS
Duration of Response (DOR) | 24 months
  Evaluate preliminary anti-tumor activity for AE071 and EVEROLIMUS
Progression Free survival (PFS) | 24 months
  Evaluate preliminary anti-tumor activity for AE071 and EVEROLIMUS
Overall Survival (OS) | 24 months
  Evaluate preliminary anti-tumor activity for AE071 and EVEROLIMUS
Concentration-time profiles of Pharmacokinetics (PK) parameters - Phase Ib | 24 months
  To characterize the PK profiles of AEB071 and EVEROLIMUS

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (3):
  - Washington University School of Medicine Dept of Oncology., St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center Onc. Dept., New York, New York
  - Sarah Cannon Research Institute Dept of Onc, Nashville, Tennessee
- Novartis Investigative Site, Rouen, France
- Germany (2):
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
- Hong Kong (2):
  - Novartis Investigative Site, New Territories, Hong Kong
  - Novartis Investigative Site, Hong Kong
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for COEB071X2103 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16288